CLINICAL TRIAL: NCT07287462
Title: Cranio-spinal Neurosurgical Approaches: Qualitative and Quantitative Analysis and Validation of New Minimally Invasive Methods on Cadaveric Anatomical Models.
Brief Title: Cranio-spinal Neurosurgical Approaches
Acronym: Neuro_SURGEM
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7155
Record Dates: First submitted 2025-11-19; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Minimally Invasive Techniques; Neurosurgical Procedures; Cadaveric Training
Keywords: Cranio-spinal surgery; Neurosurgery; Minimally invasive techniques; Surgical validation; Anatomical models; Cadaveric dissection; Neuroanatomy; Surgical training

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cranio-Spinal Neurosurgical Approaches Using Cadaveric Specimens: This cohort consists of donated human cadaveric specimens used to evaluate a range of cranio-spinal neurosurgical approaches. The group serves as an anatomical model to study surgical exposure, technical feasibility, and anatomical variation in a controlled preclinical setting. Procedures will involve macroscopic and microscopic visualization methods and may include testing of new surgical techniques or instruments. Surgeons performing the dissections will provide structured assessments of technical difficulty, visibility, and usability of the approaches.
  Interventions: Procedure: Standardized cranio-spinal neurosurgical approaches performed on donated cadaveric specimens to assess surgical exposure, feasibility, anatomical variation, and selected new techniques.

INTERVENTIONS:
Procedure: Standardized cranio-spinal neurosurgical approaches performed on donated cadaveric specimens to assess surgical exposure, feasibility, anatomical variation, and selected new techniques. — This intervention consists of performing standardized cranio-spinal neurosurgical approaches on donated human cadaveric specimens to evaluate surgical exposure, operative feasibility, and anatomical variation in a preclinical setting. The procedures use both macroscopic and microscopic visualization systems. uantitative measurements of exposure area and operative workspace are obtained through dedicated imaging and navigation-based software. The intervention also allows controlled testing of new surgical tools or techniques, with surgeon-reported assessments of difficulty, visibility, and usability. In addition, hands-on dissection sessions are incorporated to support structured surgical training and technical skill development.
  Other Names: No other names or identifiers; refers only to standardized cranio-spinal neurosurgical approaches on cadaveric specimens

SUMMARY:
The goal of this observational study is to learn how different cranio-spinal surgical approaches work and how much anatomical exposure each technique provides in donated human cadaver specimens. The study also aims to understand anatomical variations and to evaluate new surgical techniques and tools that may improve neurosurgical training and practice.

The main questions it aims to answer are:

* How much surgical exposure area and volume of work does each cranio-spinal approach allow?
* How do anatomical variations influence the effectiveness and feasibility of different approaches? Researchers will also compare results obtained using different surgical visualization methods (such as the surgical microscope approach or macroscopic evaluation) to see if any method improves visibility or operative efficiency.

Cadaveric specimens will undergo:

* Step-by-step cranio-spinal surgical approaches performed by trained neurosurgeons.
* Quantitative measurements of exposed anatomical areas using imaging software (BrainChop).
* Assessment of operative time, perceived difficulty by surgeons, and visibility of target anatomical structures.
* Testing of new surgical instruments or techniques when applicable, without involving any drugs or medical devices.

This study follows Italian regulations on post-mortem body donation for scientific research (Law No. 10/2020) and is conducted at a single research center recognized as an IRCCS (Istituto di Ricovero e Cura a Carattere Scientifico-Scientific Institute for Hospitalization and Care).

DETAILED DESCRIPTION:
This observational, monocentric, preclinical study. The main objective of this study is to conduct a systematic and quantitative preclinical analysis of multiple cranio-spinal surgical approaches, using both macroscopic and microscopic evaluation.

The study evaluates multiple surgical corridors to the cranial and spinal regions and involves detailed measurement of the volume of work and exposed anatomical area attainable with each approach. Additional technical objectives include the analysis of anatomical variations that may influence surgical execution, and the validation of new surgical techniques and instruments in a controlled laboratory environment.

All dissections will be carried out on cadaveric specimens voluntarily donated according to Italian legislation on post-mortem body donation (Law No. 10/2020). Procedures will be performed by trained neurosurgeons using standard microsurgical techniques. Quantitative measurements of exposure areas and operative volumes will be obtained using dedicated imaging software, including BrainChop.

The study also incorporates structured evaluations of technical difficulty and surgeon experience. After completing each approach, operating surgeons will provide standardized ratings of perceived difficulty, visibility of target structures, and usability of any new surgical tools or techniques tested. These assessments contribute to the systematic validation of surgical methods and instrumentation in the preclinical setting.

In addition, the study supports surgical education by integrating structured dissection sessions. Participants (surgeons or trainees) will complete pre- and post-training assessments to evaluate procedural understanding, anatomical knowledge, and perceived skill acquisition.

The study will enroll 35 cadaveric specimens over a three-year period. No drugs or implantable medical devices will be used. All specimens will be stored and handled according to institutional anatomical laboratory standards.

The statistical analysis plan includes descriptive and comparative analyses. Quantitative variables-such as exposure area, volume of work, and operative time-will be summarized as mean ± standard deviation (SD). Qualitative variables-such as visibility scores or difficulty ratings-will be reported as absolute and relative frequencies. For pre- and post-training comparisons, the paired t-test or Wilcoxon signed-rank test will be applied depending on data distribution. Comparisons of operative time or exposure metrics across techniques will be performed using Analysis of Variance (ANOVA) or the Kruskal-Wallis test. Statistical significance will be defined as p < 0.05. All analyses will be conducted using Stata statistical software (StataCorp LLC, College Station, TX, USA).

ELIGIBILITY:
Inclusion Criteria

* Cadaveric specimens from individuals who provided informed consent for post-mortem donation of their body or tissues for scientific research.
* Specimens that meet all legal requirements for anatomical donation under Italian Law No. 10/2020 and Presidential Decree (DPR) No. 47/2023.
* Specimens that are available for the full duration of the study and suitable for performing multiple cranio-spinal surgical approaches.

Exclusion Criteria

* Specimens that do not meet the legal or ethical requirements for anatomical donation as defined by Italian regulations.
* Cadavers with major anatomical deformities, advanced tissue degradation, or pathological conditions that would interfere with surgical dissection or measurement accuracy.
* Specimens lacking adequate documentation or verified donor consent for post-mortem donation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of human cadaveric specimens voluntarily donated for scientific and educational purposes under Italian post-mortem donation regulations. Specimens are obtained through the anatomical donation program of the participating institution and represent a natural range of adult anatomical variability. These cadavers serve as preclinical anatomical models for evaluating cranio-spinal neurosurgical approaches in a controlled laboratory setting. The population provides diverse anatomical characteristics that allow systematic assessment of surgical exposure, feasibility, and technical performance across different surgical corridors.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Quantification of Work Volume and Exposed Area in Cranio-Spinal Surgical Approaches | Measurements will be obtained twice for each approach on every specimen: before the dissection using baseline CT imaging and after completing the approach using repeat CT imaging on the same day.
  Work volume represents the three-dimensional operative space created by each cranio-spinal surgical approach. Quantification will be performed using BrainChop imaging software on standardized CT scans. Segmentation will follow predefined protocols to ensure reproducibility. Higher values indicate a larger and more accessible operative corridor.
  Unit of Measure: cubic millimeters (mm³).
Exposed Anatomical Surface Area Obtained by Each Surgical Approach | Measurements will be obtained twice for each approach on every specimen: before the dissection using baseline CT imaging and after completing the approach using repeat CT imaging on the same day.
  Exposed Anatomical Surface Area Obtained by Each Surgical Approach
  Description:
  Exposed area corresponds to the two-dimensional anatomical surface revealed by each surgical approach. Measurements will be obtained from CT-based reconstructions using the same standardized segmentation workflow. Higher surface values reflect wider surgical exposure.
  Unit of Measure: square millimeter

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Doglietto, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schreiber A, Ferrari M, Rampinelli V, Doglietto F, Belotti F, Lancini D, Ravanelli M, Rodella LF, Fontanella MM, Nicolai P. Modular Endoscopic Medial Maxillectomies: Quantitative Analysis of Surgical Exposure in a Preclinical Setting. World Neurosurg. 2017 Apr;100:44-55. doi: 10.1016/j.wneu.2016.12.094. Epub 2017 Jan 3. PMID 28057590
- [Background] Muhanna N, Chan H, Qiu J, Daly M, Khan T, Doglietto F, Kucharczyk W, Goldstein DP, Irish JC, de Almeida JR. Volumetric Analysis of Endoscopic and Maxillary Swing Surgical Approaches for Nasopharyngectomy. J Neurol Surg B Skull Base. 2018 Oct;79(5):466-474. doi: 10.1055/s-0037-1617432. Epub 2018 Jan 19. PMID 30210974
- [Background] Jagersberg M, Brodard J, Qiu J, Mansouri A, Doglietto F, Gentili F, Kucharczyk W, Fasel J, Schaller K, Radovanovic I. Quantification of Working Volumes, Exposure, and Target-Specific Maneuverability of the Pterional Craniotomy and Its Minimally Invasive Variants. World Neurosurg. 2017 May;101:710-717.e2. doi: 10.1016/j.wneu.2017.02.011. Epub 2017 Feb 22. PMID 28254536
- [Background] Ferrari M, Schreiber A, Mattavelli D, Lombardi D, Rampinelli V, Doglietto F, Rodella LF, Nicolai P. Surgical anatomy of the parapharyngeal space: Multiperspective, quantification-based study. Head Neck. 2019 Mar;41(3):642-656. doi: 10.1002/hed.25378. Epub 2018 Dec 28. PMID 30592348
- [Background] Ebner FH, Koerbel A, Kirschniak A, Roser F, Kaminsky J, Tatagiba M. Endoscope-assisted retrosigmoid intradural suprameatal approach to the middle fossa: anatomical and surgical considerations. Eur J Surg Oncol. 2007 Feb;33(1):109-13. doi: 10.1016/j.ejso.2006.09.036. Epub 2006 Nov 14. PMID 17110074
- [Background] Doglietto F, Belotti F, Qiu J, Roca E, Radovanovic I, Agur A, Kucharczyk W, Schreiber A, Villaret AB, Nicolai P, Gentili F, Fontanella MM. Endonasal and Transoral Approaches to the Craniovertebral Junction: A Quantitative Anatomical Study. Acta Neurochir Suppl. 2019;125:37-44. doi: 10.1007/978-3-319-62515-7_6. PMID 30610300
- [Background] Doglietto F, Qiu J, Ravichandiran M, Radovanovic I, Belotti F, Agur A, Zadeh G, Fontanella MM, Kucharczyk W, Gentili F. Quantitative comparison of cranial approaches in the anatomy laboratory: A neuronavigation based research method. World J Methodol. 2017 Dec 26;7(4):139-147. doi: 10.5662/wjm.v7.i4.139. eCollection 2017 Dec 26. PMID 29354486
- [Background] Agosti E, De Maria L, Mattogno PP, Della Pepa GM, D'Onofrio GF, Fiorindi A, Lauretti L, Olivi A, Fontanella MM, Doglietto F. Quantitative Anatomical Studies in Neurosurgery: A Systematic and Critical Review of Research Methods. Life (Basel). 2023 Aug 28;13(9):1822. doi: 10.3390/life13091822. PMID 37763226
- [Background] Liu JK, Kshettry VR, Recinos PF, Kamian K, Schlenk RP, Benzel EC. Establishing a surgical skills laboratory and dissection curriculum for neurosurgical residency training. J Neurosurg. 2015 Nov;123(5):1331-8. doi: 10.3171/2014.11.JNS14902. Epub 2015 May 26. PMID 26052729
- [Background] Bohl MA, McBryan S, Spear C, Pais D, Preul MC, Wilhelmi B, Yeskel A, Turner JD, Kakarla UK, Nakaji P. Evaluation of a Novel Surgical Skills Training Course: Are Cadavers Still the Gold Standard for Surgical Skills Training? World Neurosurg. 2019 Jul;127:63-71. doi: 10.1016/j.wneu.2019.03.230. Epub 2019 Mar 28. PMID 30930320
- [Background] Berg DA, Milner RE, Fisher CA, Goldberg AJ, Dempsey DT, Grewal H. A cost-effective approach to establishing a surgical skills laboratory. Surgery. 2007 Nov;142(5):712-21. doi: 10.1016/j.surg.2007.05.011. PMID 17981192
- [Background] Tschabitscher M, Di Ieva A. Practical guidelines for setting up an endoscopic/skull base cadaver laboratory. World Neurosurg. 2013 Feb;79(2 Suppl):S16.e1-7. doi: 10.1016/j.wneu.2011.02.045. Epub 2011 Nov 7. PMID 22120404
- [Background] Kshettry VR, Mullin JP, Schlenk R, Recinos PF, Benzel EC. The role of laboratory dissection training in neurosurgical residency: results of a national survey. World Neurosurg. 2014 Nov;82(5):554-9. doi: 10.1016/j.wneu.2014.05.028. Epub 2014 May 27. PMID 24875190
- [Background] Ghosh SK. Paying respect to human cadavers: We owe this to the first teacher in anatomy. Ann Anat. 2017 May;211:129-134. doi: 10.1016/j.aanat.2017.02.004. Epub 2017 Mar 6. PMID 28279760
- [Background] Wilkinson TM. Getting consent into perspective. Clin Anat. 2014 Sep;27(6):844-6. doi: 10.1002/ca.22412. Epub 2014 May 2. PMID 24797429
- [Background] Jones DG. Using and respecting the dead human body: an anatomist's perspective. Clin Anat. 2014 Sep;27(6):839-43. doi: 10.1002/ca.22405. Epub 2014 Apr 19. PMID 24753363
- [Background] Wilkinson TM. Respect for the dead and the ethics of anatomy. Clin Anat. 2014 Apr;27(3):286-90. doi: 10.1002/ca.22263. Epub 2013 May 29. PMID 23716492
- [Background] Larner SP, Mcquone B, Schober JM, Loukas M, Terrell M. Perceptions of the living dead: An assessment of knowledge and opinions about whole body donation, its process, and willingness to become cadaveric donors in Pennsylvania. Clin Anat. 2015 May;28(4):442-8. doi: 10.1002/ca.22516. Epub 2015 Feb 26. PMID 25727324
- [Background] McMenamin PG, McLachlan J, Wilson A, McBride JM, Pickering J, Evans DJR, Winkelmann A. Do we really need cadavers anymore to learn anatomy in undergraduate medicine? Med Teach. 2018 Oct;40(10):1020-1029. doi: 10.1080/0142159X.2018.1485884. Epub 2018 Sep 28. PMID 30265177
- [Background] Granger NA. Dissection laboratory is vital to medical gross anatomy education. Anat Rec B New Anat. 2004 Nov;281(1):6-8. doi: 10.1002/ar.b.20039. No abstract available. PMID 15558779
- [Background] McCulloch P, Altman DG, Campbell WB, Flum DR, Glasziou P, Marshall JC, Nicholl J; Balliol Collaboration; Aronson JK, Barkun JS, Blazeby JM, Boutron IC, Campbell WB, Clavien PA, Cook JA, Ergina PL, Feldman LS, Flum DR, Maddern GJ, Nicholl J, Reeves BC, Seiler CM, Strasberg SM, Meakins JL, Ashby D, Black N, Bunker J, Burton M, Campbell M, Chalkidou K, Chalmers I, de Leval M, Deeks J, Ergina PL, Grant A, Gray M, Greenhalgh R, Jenicek M, Kehoe S, Lilford R, Littlejohns P, Loke Y, Madhock R, McPherson K, Meakins J, Rothwell P, Summerskill B, Taggart D, Tekkis P, Thompson M, Treasure T, Trohler U, Vandenbroucke J. No surgical innovation without evaluation: the IDEAL recommendations. Lancet. 2009 Sep 26;374(9695):1105-12. doi: 10.1016/S0140-6736(09)61116-8. PMID 19782876

DOCUMENTS (1):
  • Study Protocol (2025-04-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT07287462/Prot_000.pdf